CLINICAL TRIAL: NCT00503984
Title: A Phase I/II Study of Azacitidine (Vidaza), Docetaxel and Prednisone for Patients With Hormone Refractory Metastatic Prostate Cancer Previously Treated With a Taxotere Containing Regimen.
Brief Title: A Phase I/II Study of Azacitidine, Docetaxel, and Prednisone for Metastatic Prostate Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of Funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Rakesh Singal, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061143; SCCC-2006080 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20070344 (Other: Western Institutional Review Board); 20140376 (Other: University of Miami)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer; Pain
Keywords: Adenocarcinoma of the prostate; Recurrent prostate cancer; Stage IV prostate cancer; Pain
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — Azacitidine; Docetaxel; Prednisone; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 - Aza + Doc (Experimental): Phase 1 Azacitidine (Aza) and Docetaxel (Doc) with dose escalation/de-escalation design, and Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim).
  Interventions: Drug: Azacitidine; Drug: Docetaxel; Drug: Prednisone; Genetic: GADD45α methylation and expression analysis; Drug: Pegfilgrastim; Drug: Filgrastim
- Phase 2 - Aza + Doc RPTD (Experimental): Recommended Phase Two Dose (RPTD) of Azacitidine and Docetaxel; and Prednisone; with optional growth factor support (pegfilgrastim/filgrastim).
  Interventions: Drug: Azacitidine; Drug: Docetaxel; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Filgrastim

INTERVENTIONS:
Drug: Azacitidine — Intravenous infusion over 30 minutes Days 1 - 5 of each 3 weekly cycle.
  Other Names: Vidaza®
Drug: Docetaxel — Intravenous infusion over 1 hour on day 6 of each 3 weekly cycle.
  Other Names: Taxotere®
Drug: Prednisone — Patient will receive prednisone 5mg twice a day from Day 1 to 21 of each cycle.
Genetic: GADD45α methylation and expression analysis — Peripheral blood samples from patients will be collected as described in section 8.1 (total of 4 blood samples). DNA will be isolated from serum, bisulfite treated and evaluated for methylation by bisulfite genomic sequencing.
  Patients with accessible prostate tissue or metastases will undergo biopsy prior to treatment if they consent to do so.
  Arms: Phase 1 - Aza + Doc
Drug: Pegfilgrastim — Growth factor support.Granulocyte-colony stimulating factor (G-CSF)
  Other Names: Neulasta
Drug: Filgrastim — Growth factor support. Granulocyte-colony stimulating factor (G-CSF)
  Other Names: Neupogen

SUMMARY:
Azacitidine can reverse clinical resistance to docetaxel through upregulation of Growth Arrest and DNA Damage inducible alpha (GADD45α) and other epigenetically regulated genes.

DETAILED DESCRIPTION:
Study design A phase I/II clinical trial in patients with hormone refractory metastatic prostate cancer.

Primary objective phase I component of study:

To determine a safe and potentially efficacious phase II dose of azacitidine in combination with docetaxel and prednisone that can be used for the treatment of hormone refractory metastatic prostate cancer.

Primary objective phase II component of study:

To determine the therapeutic efficacy of combined therapy of azacitidine, docetaxel, and prednisone, in the treatment of hormone refractory metastatic prostate cancer. The primary measure of therapeutic efficacy is response, defined as prostate-specific antigen (PSA) response, complete response (CR), or partial response (PR).

Secondary endpoints are toxicity, duration of response, progression-free survival, and overall survival.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient who had histologically confirmed adenocarcinoma of the prostate.
* Patient must have radiologically documented metastatic disease.
* Patients should have received at least 12 weeks of docetaxel chemotherapy or a cumulative docetaxel dose of 300 mg/m2 and have disease progression on docetaxel-based therapy. Patients must have progressed after prior hormonal therapy (e.g. medical or surgical castration) as defined by a castrate level of testosterone (less than 50 ng/mL). If patient underwent medical castration, it must be continued during the study.
* Progressive disease may be documented by:

  * Non-measurable disease:

    * Serum PSA progression defined as a rise in at least 2 consecutive serum PSA values, each obtained at least 1 week apart and an absolute value greater than 2.0 ng/ml or,
    * Appearance of two or more new lesions on bone scan.
    * Patients with treated epidural lesions and no other epidural progression will be eligible.
  * Measurable disease

    * Documented progression of disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria demonstrating at least one visceral or soft tissue metastatic lesion (including new lesion).
    * Nodal or visceral progression will be sufficient for trial entry independent of PSA
    * Only lymph nodes ≥ 2 cm in diameter will be used to assess for a change in size.
    * Previously irradiated lesions, primary prostatic lesion, and bone lesions will be considered non-measurable disease.
* Patient is 18 years or older.
* Patient had a Karnofsky Performance Status (KPS) of at least 70% or Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2.
* Life expectancy of > 6 months.
* Patient with adequate organ function as defined as

  * Absolute Neutrophils Count greater than 1500 cells/mm3
  * Platelets greater than 100,000 cells/mm3
  * Hemoglobin greater than 8 g/dL,
  * Adequate liver function as documented by:

    * Total Bilirubin </= 1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
    * AST and ALT </= 2.5 ULN. (In determining eligibility the more abnormal of the two values (AST or ALT) should be used.)
  * Serum creatinine </= 2.0 mg/dl or </= 1.5 x institutional upper limit of normal.
* Male patient must be willing to use an acceptable barrier method for contraception; and must agree not to father a child whilst receiving treatment with Azacitidine and up to six months after last dose.
* Patients may have a history of prior malignancy (≥ 5 years prior) provided that the patient is currently disease free and off all therapy for that malignancy. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patients must be informed of the investigational nature of the treatment and must give signed written and informed consent.

EXCLUSION CRITERIA:

* Patients who have received strontium 89 (metastron®), Samarium 153 (quadramet®) radiation therapy within 8 weeks of enrollment.
* Evidence of significant active infection during screening for eligibility.
* Patients who have had a psychiatric illness that could potentially interfere with completion of treatment according to protocol.
* Patients who had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. There is no wash-out period for patients who received Zytiga.
* Patient who had brain metastases.
* Patient who had history of allergic reactions attributed to compound or similar chemical or biological composition to azacitidine (Vidaza®) or docetaxel or other drugs formulated with polysorbate 80 or mannitol.
* Patient had major surgical procedure within 28 days before Day 1 of treatment.
* Hepatic malignancy.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Singal, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Background] Singal R, Ramachandran K, Gordian E, Quintero C, Zhao W, Reis IM. Phase I/II study of azacitidine, docetaxel, and prednisone in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel-based therapy. Clin Genitourin Cancer. 2015 Feb;13(1):22-31. doi: 10.1016/j.clgc.2014.07.008. Epub 2014 Aug 1. PMID 25178642

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Level 1 - 75 Aza + 60 Doc: All Phase 1 participants who received at least one dose starting at the Level 1 dose combination of 75 mg/m^2 of Azacitidine (Aza), 60 mg/m^2 of Docetaxel (Doc) and 5mg of Prednisone.
- Phase 1: Level 2 - 75 Aza + 75 Doc: All Phase 1 participants who received at least one dose starting at the Level 2 dose combination of 75 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) and 5mg of Prednisone.
- Phase 1: Level 3 - 100 Aza + 75 Doc: All Phase 1 participants who received at least one dose starting at the Level 3 dose combination of 100 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) and 5mg of Prednisone.
- Phase 1: Level 4 - 150 Aza + 75 Doc: All Phase 1 participants who received at least one dose starting at the Level 4 dose combination of 150 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) and 5 mg of Prednisone.
- Phase 2 - Aza + Doc Initial RPTD: All Phase 2 participants who received at least one dose of the combination of Azacitidine and Docetaxel with 5 mg of Prednisone at the recommended phase two dose level (RPTD).
- Phase 2 - Aza + Doc Reduced RPTD: All Phase 2 participants who received at least one reduced dose of the combination of Azacitidine and Docetaxel with 5 mg of Prednisone at the recommended phase two dose level (RPTD).
Period: Overall Study
Arm/Group | Phase 1: Level 1 - 75 Aza + 60 Doc | Phase 1: Level 2 - 75 Aza + 75 Doc | Phase 1: Level 3 - 100 Aza + 75 Doc | Phase 1: Level 4 - 150 Aza + 75 Doc | Phase 2 - Aza + Doc Initial RPTD | Phase 2 - Aza + Doc Reduced RPTD
Started | 3 | 3 | 3 | 6 | 6 | 1
Completed | 3 | 1 | 3 | 6 | 5 | 1
Not Completed | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: All Phase 1 participants who received at least one dose of the combination of Azacitidine (Aza) and Docetaxel (Doc) and 5mg of Prednisone at one of the starting dose levels:
  * Level 1: 75 mg/m2 Aza + 60 mg/m2 Doc
  * Level 2: 75 mg/m2 Aza + 75 mg/m2 Doc
  * Level 3: 100 mg/m2 Aza + 75 mg/m2 Doc
  * Level 4: 150 mg/m2 Aza + 75 mg/m2 Doc
- Phase 2: All Phase 2 participants who received at least one dose of the combination of Azacitidine and Docetaxel with 5 mg of Prednisone at the recommended phase two dose level (RPTD).
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Customized [Number; unit: participants]
  < 60 years | 3 | 1 | 4
  60 - 69 years | 8 | 3 | 11
  >= 70 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Recommended Phase Two Dose (RPTD) of Azacitidine and Docetaxel in Combination With Prednisone. (Azacitidine and Docetaxel)
Description: Determination of a safe and potentially efficacious phase II dose of azacitidine in combination with docetaxel and prednisone that can be used for the treatment of hormone refractory metastatic prostate cancer.
Time Frame: Up to 1.5 years
Population: Number of participants enrolled in the Phase 1 portion of the study. The initial RPTD was 150 mg/m2 Azacitidine + 75 mg/m2 Docetaxel, with 5mg of Prednisone. However, due to the death of one patient, the Data and Safety Monitoring Board (DSMB) recommended that the RPTD be reduced to 75 mg/m2 Azacitidine + 75 mg/m2 Docetaxel, with 5mg of Prednisone.
Measure: Number; unit: mg/m2
Arm/Group | Phase 1 - Aza + Doc
Number analyzed (Participants) | 15
mg/m2
  Initial RPTD Azacitidine (mg/m2) | 150
  Initial RPTD Docetaxel (mg/m2) | 75
  Reduced RPTD Azacitidine (mg/m2) | 75
  Reduced RPTD Docetaxel (mg/m2) | 75

2. Primary Outcome: Phase I - Recommended Phase Two Dose (RPTD) of Azacitidine and Docetaxel in Combination With Prednisone. (Prednisone)
Description: as for outcome 1
Time Frame: Up to 1.5 years
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Phase 1 - Aza + Doc
Number analyzed (Participants) | 15
mg
  Initial RPTD Prednisone (mg) | 5
  Reduced RPTD Prednisone (mg) | 5

3. Primary Outcome: Number of Participants Achieving Prostate-specific Antigen (PSA) Response.
Description: Number of participants achieving prostate-specific antigen (PSA) response according to Prostate Cancer Working Group 1 (PCWG1) criteria. PSA response according to PCWG1 is defined as an least 50 percent decline in PSA level from baseline that was maintained for at least three weeks.
Time Frame: Up to 4.5 years.
Population: Of the 22 participants enrolled, only 19 were evaluable because they completed 2 or more cycles of protocol therapy.
Measure: Number; unit: participants
Groups:
- Phase 1: Level 1 - 75 Aza + 60 Doc: Phase 1, Starting Dose Level 1: 75 mg/m^2 of Azacitidine (Aza), 60 mg/m^2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 2 - 75 Aza + 75 Doc: Phase 1, Starting Dose Level 2: 75 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 3 - 100 Aza + 75 Doc: Phase 1, Starting Dose Level 3: 100 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 4 - 150 Aza + 75 Doc: Phase 1, Starting Dose Level 1: 150 mg/m^2 of Azacitidine (Aza), 75 mg/m^2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 2 - Aza + Doc Initial RPTD: Recommended Phase Two Dose (RPTD) of Azacitidine and Docetaxel; and Prednisone; with optional growth factor support (pegfilgrastim/filgrastim).
Arm/Group | Phase 1: Level 1 - 75 Aza + 60 Doc | Phase 1: Level 2 - 75 Aza + 75 Doc | Phase 1: Level 3 - 100 Aza + 75 Doc | Phase 1: Level 4 - 150 Aza + 75 Doc | Phase 2 - Aza + Doc Initial RPTD | Phase 2 - Aza + Doc Reduced RPTD
Number analyzed (Participants) | 3 | 1 | 3 | 6 | 5 | 1
participants | 0 | 1 | 2 | 4 | 3 | 0

4. Primary Outcome: Number of Participants Achieving Complete Response (CR) or Partial Response (CR) to Protocol Therapy.
Description: Number of participants achieving Complete Response (CR) or Partial Response to protocol therapy according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.0 Criteria. Per RECIST 1.0 for target lesions and assessed by MRI: "Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; "
Time Frame: Up to 4.5 years
Population: Number of evaluable participants with measurable disease on CT scan. Only 10 of the 19 evaluable participants had measurable disease on CT Scan.
Measure: Number; unit: participants
Groups:
- Phase 1: Level 1 - 75 Aza + 60 Doc: Phase 1, Starting Dose Level 1: 75 mg/m2 of Azacitidine (Aza), 60 mg/m2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 2 - 75 Aza + 75 Doc: Phase 1, Starting Dose Level 2: 75 mg/m2 of Azacitidine (Aza), 75 mg/m2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 3 - 100 Aza + 75 Doc: Phase 1, Starting Dose Level 3: 100 mg/m2 of Azacitidine (Aza), 75 mg/m2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 1: Level 4 - 150 Aza + 75 Doc: Phase 1, Starting Dose Level 4: 150 mg/m2 of Azacitidine (Aza), 75 mg/m2 of Docetaxel (Doc) with dose escalation/de-escalation design, and 5 mg of Prednisone, with growth factor support; GADD45α methylation and expression analysis, with optional growth factor support (pegfilgrastim/filgrastim)
- Phase 2 - Aza + Doc Initial RPTD: Initial Recommended Phase Two Dose (RPTD) of Azacitidine and Docetaxel; and Prednisone; with optional growth factor support (pegfilgrastim/filgrastim).
Arm/Group | Phase 1: Level 1 - 75 Aza + 60 Doc | Phase 1: Level 2 - 75 Aza + 75 Doc | Phase 1: Level 3 - 100 Aza + 75 Doc | Phase 1: Level 4 - 150 Aza + 75 Doc | Phase 2 - Aza + Doc Initial RPTD
Number analyzed (Participants) | 2 | 0 | 2 | 3 | 3
participants
  Complete Response (CR) | 0 |  | 1 | 0 | 0
  Partial Response (PR) | 0 |  | 0 | 1 | 1

5. Secondary Outcome: Duration of Response
Description: Length of time from the date of first observation of complete response (CR) or partial response (PR) to the date of first observation of disease progression, according to prostate-specific antigen (PSA) response according to Prostate Cancer Working Group 1 (PCWG1) criteria. PSA response according to PCWG1 is defined as an least 50 percent decline in PSA level from baseline that was maintained for at least three weeks.
Time Frame: Up to 4.5 years.
Population: The 10 participants in both Phase 1 and Phase 2 who achieved PSA response.
Measure: Median (Full Range); unit: weeks
Groups:
- All Study Participants Achieving PSA Response: All study participants who achieved PSA response to protocol therapy. PSA response according to PCWG1 is defined as an least 50 percent decline in PSA level from baseline that was maintained for at least three weeks.
Arm/Group | All Study Participants Achieving PSA Response
Number analyzed (Participants) | 10
weeks | 20.5 [3 to 63.4]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: The time from the date of start of treatment until the first documented or confirmed disease progression, or death related to prostate cancer, whichever is earlier.
Time Frame: Up to 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Study Participants: All study participants who received at least one dose of combination Azacitidine + Docetaxel, and 5 mg of Prednisone in either Phase 1 or Phase 2.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
months | 4.9 [1.4 to 9.5]

7. Secondary Outcome: Overall Survival (OS)
Description: The time from the date of initiation of study treatment until date of death from any cause.
Time Frame: Up to 4.5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
months | 19.5 [13.6 to 26.4]

8. Secondary Outcome: Number of Participants Experiencing Adverse Events After Beginning Protocol Therapy.
Time Frame: Up to 4.5 years
Population: All study participants who received at least one dose of combination Azacitidine + Docetaxel, and 5 mg of Prednisone in either Phase 1 or Phase 2.
Measure: Number; unit: participants
Groups:
- Level 1 - 75 Aza + 60 Doc: 75 mg/m2 of Azacitidine (Aza) and 60 mg/m2 of Docetaxel (Doc)
- Level 2 - 75 Aza + 75 Doc: 75 mg/m2 of Azacitidine (Aza) and 75 mg/m2 of Docetaxel (Doc)
- Level 3 - 100 Aza + 75 Doc: 100 mg/m2 of Azacitidine (Aza) and 75 mg/m2 of Docetaxel (Doc)
- Level 4 - 150 Aza + 75 Doc: 150 mg/m2 of Azacitidine (Aza) and 75 mg/m2 of Docetaxel (Doc)
Arm/Group | Level 1 - 75 Aza + 60 Doc | Level 2 - 75 Aza + 75 Doc | Level 3 - 100 Aza + 75 Doc | Level 4 - 150 Aza + 75 Doc
Number analyzed (Participants) | 3 | 4 | 3 | 12
participants | 3 | 4 | 3 | 12

ADVERSE EVENTS:
Description: All Phase 1 and Phase 2 participants
Arm/Group | Level 1 - 75 Aza + 60 Doc | Level 2 - 75 Aza + 75 Doc | Level 3 - 100 Aza + 75 Doc | Level 4 - 150 Aza + 75 Doc
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 1/3 | 4/12
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 - 75 Aza + 60 Doc (N=3) | Level 2 - 75 Aza + 75 Doc (N=4) | Level 3 - 100 Aza + 75 Doc (N=3) | Level 4 - 150 Aza + 75 Doc (N=12)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Infection, normal ANC, Catheter-related (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 - 75 Aza + 60 Doc (N=3) | Level 2 - 75 Aza + 75 Doc (N=4) | Level 3 - 100 Aza + 75 Doc (N=3) | Level 4 - 150 Aza + 75 Doc (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (62)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (10) | 2 (9) | 4 (51)
Leukocytes (Blood and lymphatic system disorders) | 1 (3) | 2 (19) | 3 (12) | 8 (72)
Neutrophils (Blood and lymphatic system disorders) | 3 (5) | 2 (10) | 3 (7) | 6 (31)
Platelets (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (13)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (9)
Fatigue (General disorders) | 2 (3) | 1 (3) | 3 (3) | 8 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 2 (4) | 3 (18)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Back Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (6)
Allergic reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (10)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Edema limbs (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Weight loss (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (11)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy - Other (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (5) | 2 (2) | 7 (9)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection Site Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Musculosketal - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rigors/Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes